CLINICAL TRIAL: NCT00933153
Title: Validation of the Malnutrition Screening Tool (MST) and Effectiveness of Oral Nutritional Supplements (ONS) on Weight, Nutritional Status and Quality of Life in a Meals-on-Wheels Population
Brief Title: Effectiveness of Oral Nutritional Supplements (ONS) in a Meals-on-Wheels Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Gina Hill, Associate Professor, Texas Christian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCUMOW1
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Elderly; Malnutrition
Keywords: Elderly; Malnutrition; Oral Nutrition Supplement; Meals on Wheels
MeSH Terms: conditions — Malnutrition | interventions — Ensure Plus; Food Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meals on Wheels (Active Comparator): Participants will receive two meals daily from Meals on Wheels.
  Interventions: Dietary Supplement: Meals on Wheels
- Meals on Wheels + Ensure Plus supplement (Experimental): Participants will receive two meals from Meals on Wheels daily plus Ensure Plus supplements with meals.
  Interventions: Dietary Supplement: Ensure Plus; Dietary Supplement: Meals on Wheels

INTERVENTIONS:
Dietary Supplement: Ensure Plus — Ensure plus supplement with meals
  Arms: Meals on Wheels + Ensure Plus supplement
Dietary Supplement: Meals on Wheels — Two Meals on Wheels twice daily

SUMMARY:
Researchers will measure weight, height, hand grip strength and quality of life information of Meals on Wheels (MOW) clients who are considered to have nutrition problems. Participants will randomly be put into a group that receives either typical meals from Meals on Wheels or Ensure Plus supplements with their meals. Three months later the same data will be collected again. The objective of this study is to demonstrate the effectiveness of providing oral nutritional supplements (ONS) to MOW clients with or at risk of malnutrition on nutritional status over a 3-month period.

DETAILED DESCRIPTION:
While it is well known that older adults are at increased nutritional risk and that nutrition intervention, such as oral nutritional supplementation (ONS) is beneficial in this population, there is limited research on the effect of oral nutritional supplements (ONS) in the Meals on Wheels population. This prospective randomized controlled trial will determine the effectiveness of oral nutritional supplements (ONS) in addition to daily meals from Meals on Wheels on weight status, hand grip strength, quality of life, and malnutrition screening scores in MOW clients with or at-risk of malnutrition over a 3-month study period.

ELIGIBILITY:
Inclusion Criteria:

* Participant is Meals on Wheels Inc. of Tarrant County client.
* Participant is 60 years of age or older.
* Participant is identified as medium or high risk of malnutrition as defined by the MST (Medium Risk MST score =2-3 or High Risk MST score =4-5).
* Participant is willing and/or able to consume oral nutritional supplements (ONS).
* Participant provides written informed consent to participate in the study.
* Participant provides authorization to use and/or disclose personal and/or health data.

Exclusion Criteria:

* Patient cannot safely consume an oral nutritional supplement (ONS).

  * Example Patient has active gastrointestinal disease (e.g., intestinal obstruction, inflammatory bowel disease, ischemic colitis, diverticulitis, irritable bowel disease, pancreatitis).
* Patient has Diabetes mellitus.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina J Hill, PhD, Principal Investigator — Texas Christian University; Sherry Simon, BS, Study Director — Meals on Wheels Inc. of Tarrant County
Locations (1):
- Meals on Wheels, Inc. of Tarrant County, Fort Worth, Texas, United States

REFERENCES:
- See also: Texas Christian University — http://www.tcu.edu
- See also: Meals on Wheels Inc. Tarrant County — http://www.mealsonwheels.org